CLINICAL TRIAL: NCT06626971
Title: A Phase II Clinical Trial on the Use of ARA 290 for the Treatment of Diabetic Macular Oedema
Brief Title: The Use of ARA290 for the Treatment of Diabetic Macular Oedema
Acronym: ARA290DMO
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Expiry of study drug - no replacement available.
Sponsor: Belfast Health and Social Care Trust (Other)
Collaborators: Araim Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14166NL-AS
Record Dates: First submitted 2018-03-28; First posted 2024-10-04 (Actual); Last update posted 2024-10-04 (Actual); Status verified 2024-06

CONDITIONS: Diabetic Macular Oedema
MeSH Terms: interventions — cibinetide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Intervention (Other): Subcutaneous daily injection of ARA 290 at a dose of 4mg for 12 weeks.
  Interventions: Drug: ARA290

INTERVENTIONS:
Drug: ARA290 — 4 mg subcutaneous injections of ARA290 over an 84 day period
  Other Names: L-Pyroglutamyl-L-glutamyl-L-glutaminyl-L-leucyl-L-glutamyl-L-arginyl-L-alanyl-L-leucyl-L-asparaginyl-L-seryl-L-serine

SUMMARY:
ARA 290-DMO is a prospective, open label, interventional, single centre, investigator led, phase II trial to examine the effect of ARA 290 on diabetic macular oedema in patients with type 1 or 2 diabetes.

The aim or primary objective of the study was to determine whether ARA 290 administered at a daily dose of 4mg subcutaneously for 12 weeks to patients with diabetes mellitus (DM) and DMO would have a beneficial effect on mean change in best corrected visual acuity (BCVA) from baseline values to week 12.

DETAILED DESCRIPTION:
Diabetic retinopathy a very most common cause of sight loss in people of working age. Sight loss occurs in diabetes because of diabetic macular oedema (DMO) and/or proliferative diabetic retinopathy (PDR), both are complications of diabetes in the eye.

In DMO fluid accumulates in the macula, the area responsible for our central sight. As the fluid accumulates the sight drops. The current treatments for DMO include laser and anti VEGF drugs and steroids. Anti VEGF drugs have been very helpful in the treatment of DMO. However, anti VEGF drugs need to be given by an injection into the eye, an Ophthalmologist (eye specialist) or a specialist nurse (a nurse trained for this purpose) will need to deliver this treatment to patients with DMO in the hospital.

Furthermore, patients require injections every four weeks during the first months of treatment and long term treatment is required. Moreover, not all patients respond to anti VEGFs: In 40% of patients the sight may not improve despite these injections. Because many patients with DMO have DMO in both eyes, injections need to be given in both eyes to many patients.

Given the above facts there appeared a clear need to develop new treatments for people with DMO. ARA 290 is a drug that has marked anti-inflammatory properties and has an effect in preventing the death of cells. As inflammation is known to play a role in the occurrence of DMO, it was thought that ARA 290 could potentially be helpful in treating patients with this condition. In light of this, the Investigators carried out this study to find out if ARA 290 was effective in drying the fluid in DMO. If this treatment was successful, benefits may have included a reduction of the demands on health care services and patient benefits of: self administration of the drug at home by the patients; a reduction in hospital visits; treatment of both eyes at once, reduced risks associated with injections; a more pleasant treatment (subcutaneous injection versus an injection into the eye).

ELIGIBILITY:
Inclusion Criteria:

1. Patients with DR and centre involving DMO with a central subfield thickness of > 400 microns, as determined using SD-OCT;
2. >= 18 years of age
3. Clear media and naïve to previous treatments for DMO.

Exclusion Criteria:

1. Macular oedema related to other retinal disease
2. Hazy media that prevents adequate retinal imaging
3. Allergy to fluorescein
4. Previous treatments for DMO
5. DMO with central subfield thickness of < 400 microns
6. Patients on systemic or topical steroids
7. Use of erythropoiesis stimulating agents within the two months prior to screening or during the trial
8. Treated with any other investigational medication or device within 60 days
9. Pregnant women, women who have not yet reached the menopause (no menses for 12 months or more without an alternative medical cause) who test positive for pregnancy or who are unwilling to take a pregnancy test prior to trial entry or are unwilling to undertake adequate precautions to prevent pregnancy for the duration of the trial.
10. Men who have a female partner and who are unwilling to undertake adequate precautions to prevent pregnancy for the duration of the trial.
11. Female patients who are breastfeeding
12. Active proliferative diabetic retinopathy (PDR) requiring treatment.
13. Patients with other eye diseases besides DR
14. Patients who are unable or unwilling to commit to the study schedule of events
15. Serious illness that is likely to affect the patient's ability to complete the study

Any patient showing a clinically significant improvement between the initial screening and presenting for the first screening/baseline visit may no longer be eligible for the study and will be recorded as a screen failure and will not be entered on to the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2017-05-12 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Primary Outcome - Best corrected distance visual acuity. | From baseline to week 12 (+/- 7 days)
  Best corrected distance visual acuity will be obtained in both eyes by a trained optometrist using the Early Treatment Diabetic Retinopathy Study (ETDRS) charts at baseline and at week 12. The EDTRS total score will be recorded and used for the analysis.

SECONDARY OUTCOMES:
Secondary Outcome - Central subfield thickness | Changes from baseline to week 12 (+/- 7 days).
  Central subfield retinal thickness (CST), as obtained in the central 1 mm area, will be determined by spectral domain optical coherence tomography (SD-OCT) and used for the analysis.
Secondary Outcome - Central retinal sensitivity | Changes from baseline to week 12 (+/- 7 days)
  Retinal sensitivity will be determined by macular microperimetry in both eyes.
Secondary Outcome - Retinal perfusion | Changes from baseline to week 12 (+/- 7 days)
  Retinal perfusion will be assessed by wide angle fundus fluorescein angiography (FFA).
Secondary Outcome - Tear production | Changes from baseline to week 12 (+/- 7 days)
  The Schirmer test will be performed to measure tear production.
Secondary Outcome - Patient reported outcome | Changes from baseline to week 12 (+/- 7 days)
  Patient reported outcomes will be evaluated by means of EQ-5D 5L questionnaires which will be administered to patients at baseline and at week 12 (and at week 16 if applicable).
Secondary Outcome - Change in inflammatory markers | Changes from baseline to week 12 (+/- 7 days)
  A blood sample will be used to test for ARA 290 antibodies and to complete an exploratory analysis to determine levels of inflammatory markers and carbamylated and glycosylated albumin.
Secondary Outcome - Number of Adverse events | Changes from baseline to week 12 (+/- 7 days)
  Adverse events
Secondary Outcome -% of participants with ≥ 15 ETDRS letter gain | baseline to week 12
  using Best corrected distance visual acuity
Secondary Outcome -% of participants with ≥ 10 ETDRS letter gain | baseline to week 12
  using Best corrected distance visual acuity
Secondary Outcome - Patient reported outcomes | Changes from baseline to week 12 (+/- 7 days)
  Patient reported outcomes will be evaluated by means of NEI VFQ-25 questionnaires which will be administered to patients at baseline and at week 12 (and at week 16 if applicable).
Secondary Outcome - Change in glycosylated albumin | Changes from baseline to week 12 (+/- 7 days)
  A blood sample will be used to test for ARA 290 antibodies and to complete an exploratory analysis to determine levels of inflammatory markers and carbamylated and glycosylated albumin.
Secondary Outcome - Change in carbamylated albumin | Changes from baseline to week 12 (+/- 7 days)
  A blood sample will be used to test for ARA 290 antibodies and to complete an exploratory analysis to determine levels of inflammatory markers and carbamylated and glycosylated albumin.

OTHER OUTCOMES:
Exploratory Outcome - Change in Adenosine Deaminase (ADA) | Baseline to week 12 (+/- 7 days)
  Inflammatory markers will be evaluated to investigate the potential anti-inflammatory effect of this treatment.
Exploratory Outcome - Change in Artemin (ARTN) | Baseline to week 12 (+/- 7 days)
  Inflammatory markers will be evaluated to investigate the potential anti-inflammatory effect of this treatment.
Exploratory Outcome - Axin-1 (AXIN1) | Baseline to week 12 (+/- 7 days)
  Inflammatory markers will be evaluated to investigate the potential anti-inflammatory effect of this treatment.
Exploratory Outcome - Beta-nerve growth factor (BDNF) | Baseline to week 12 (+/- 7 days)
  Inflammatory markers will be evaluated to investigate the potential anti-inflammatory effect of this treatment.
Exploratory Outcome - Caspase 8 (CASP-8) | Baseline to week 12 (+/- 7 days)
  Inflammatory markers will be evaluated to investigate the potential anti-inflammatory effect of this treatment.
Exploratory Outcome - C-C motif chemokine 4 (CCL4) | Baseline to week 12 (+/- 7 days)
  Inflammatory markers will be evaluated to investigate the potential anti-inflammatory effect of this treatment.
Exploratory Outcome - C-C motif chemokine 19 (CCL19) | Baseline to week 12 (+/- 7 days)
  Inflammatory markers will be evaluated to investigate the potential anti-inflammatory effect of this treatment.
Exploratory Outcome - C-C motif chemokine 20 (CCL20) | Baseline to week 12 (+/- 7 days)
  Inflammatory markers will be evaluated to investigate the potential anti-inflammatory effect of this treatment.
Exploratory Outcome - C-C motif chemokine 25 (CCL25) | Baseline to week 12 (+/- 7 days)
  Inflammatory markers will be evaluated to investigate the potential anti-inflammatory effect of this treatment.
Exploratory Outcome - C-C motif chemokine 28 (CCL28) | Baseline to week 12 (+/- 7 days)
  Inflammatory markers will be evaluated to investigate the potential anti-inflammatory effect of this treatment.
Exploratory Outcome - CD40L receptor (CD40) | Baseline to week 12 (+/- 7 days)
  Inflammatory markers will be evaluated to investigate the potential anti-inflammatory effect of this treatment.
Exploratory Outcome - CUB domain-containing protein 1 (CDCP1) | Baseline to week 12 (+/- 7 days)
  Inflammatory markers will be evaluated to investigate the potential anti-inflammatory effect of this treatment.
Exploratory Outcome - C-X-C motif chemokine 1 (CXCL1) | Baseline to week 12 (+/- 7 days)
  Inflammatory markers will be evaluated to investigate the potential anti-inflammatory effect of this treatment.
Exploratory Outcome - C-X-C motif chemokine 5 (CXCL5) | Baseline to week 12 (+/- 7 days)
  Inflammatory markers will be evaluated to investigate the potential anti-inflammatory effect of this treatment.
Exploratory Outcome -C-X-C motif chemokine 6 (CXCL6) | Baseline to week 12 (+/- 7 days)
  Inflammatory markers will be evaluated to investigate the potential anti-inflammatory effect of this treatment.
Exploratory Outcome -C-X-C motif chemokine 9 (CXCL9) | Baseline to week 12 (+/- 7 days)
  Inflammatory markers will be evaluated to investigate the potential anti-inflammatory effect of this treatment.
Exploratory Outcome -C-X-C motif chemokine 10 (CXCL10) | Baseline to week 12 (+/- 7 days)
  Inflammatory markers will be evaluated to investigate the potential anti-inflammatory effect of this treatment.
Exploratory Outcome -C-X-C motif chemokine 11 (CXCL11) | Baseline to week 12 (+/- 7 days)
  Inflammatory markers will be evaluated to investigate the potential anti-inflammatory effect of this treatment.
Exploratory Outcome -Cystatin D (CST5) | Baseline to week 12 (+/- 7 days)
  Inflammatory markers will be evaluated to investigate the potential anti-inflammatory effect of this treatment.
Exploratory Outcome -Delta and Notch-like epidermal growth factor related recep (DNER) | Baseline to week 12 (+/- 7 days)
  Inflammatory markers will be evaluated to investigate the potential anti-inflammatory effect of this treatment.
Exploratory Outcome -Eotaxin-1 (CCL11) | Baseline to week 12 (+/- 7 days)
  Inflammatory markers will be evaluated to investigate the potential anti-inflammatory effect of this treatment.
Exploratory Outcome -karyotic translation initiation factor 4Ebinding protein 1 (4E-BP1) | Baseline to week 12 (+/- 7 days)
  Inflammatory markers will be evaluated to investigate the potential anti-inflammatory effect of this treatment.
Exploratory Outcome -Fibroblast growth factor 5 (FGF-5) | Baseline to week 12 (+/- 7 days)
  Inflammatory markers will be evaluated to investigate the potential anti-inflammatory effect of this treatment.
Exploratory Outcome -Fibroblast growth factor 19 (FGF-19) | Baseline to week 12 (+/- 7 days)
  Inflammatory markers will be evaluated to investigate the potential anti-inflammatory effect of this treatment.
Exploratory Outcome -Fibroblast growth factor 21 (FGF-21) | Baseline to week 12 (+/- 7 days)
  Inflammatory markers will be evaluated to investigate the potential anti-inflammatory effect of this treatment.
Exploratory Outcome -Fibroblast growth factor 23 (FGF-23) | Baseline to week 12 (+/- 7 days)
  Inflammatory markers will be evaluated to investigate the potential anti-inflammatory effect of this treatment.
Exploratory Outcome -Fms-related tyrosine kinase 3 ligand (Flt3L) | Baseline to week 12 (+/- 7 days)
  Inflammatory markers will be evaluated to investigate the potential anti-inflammatory effect of this treatment.
Exploratory Outcome -Fractalkine (CX3CL1) | Baseline to week 12 (+/- 7 days)
  Inflammatory markers will be evaluated to investigate the potential anti-inflammatory effect of this treatment.
Exploratory Outcome -Glial cell line-derived neurotrophic factor (hGDNF) | Baseline to week 12 (+/- 7 days)
  Inflammatory markers will be evaluated to investigate the potential anti-inflammatory effect of this treatment.
Exploratory Outcome -Hepatocyte growth factor (HGF) | Baseline to week 12 (+/- 7 days)
  Inflammatory markers will be evaluated to investigate the potential anti-inflammatory effect of this treatment.
Exploratory Outcome -Interferon gamma (IFN-gamma) | Baseline to week 12 (+/- 7 days)
  Inflammatory markers will be evaluated to investigate the potential anti-inflammatory effect of this treatment.
Exploratory Outcome -Interleukin-1 alpha (IL-1 alpha) | Baseline to week 12 (+/- 7 days)
  Inflammatory markers will be evaluated to investigate the potential anti-inflammatory effect of this treatment.
Exploratory Outcome -Interleukin-2 (IL-2) | Baseline to week 12 (+/- 7 days)
  Inflammatory markers will be evaluated to investigate the potential anti-inflammatory effect of this treatment.
Exploratory Outcome -Interleukin-2 receptor subunit beta (IL-2RB) | Baseline to week 12 (+/- 7 days)
  Inflammatory markers will be evaluated to investigate the potential anti-inflammatory effect of this treatment.
Exploratory Outcome -Interleukin-4 (IL-4) | Baseline to week 12 (+/- 7 days)
  Inflammatory markers will be evaluated to investigate the potential anti-inflammatory effect of this treatment.
Exploratory Outcome -Interleukin-5 (IL-5) | Baseline to week 12 (+/- 7 days)
  Inflammatory markers will be evaluated to investigate the potential anti-inflammatory effect of this treatment.
Exploratory Outcome -Interleukin-6 (IL-6) | Baseline to week 12 (+/- 7 days)
  Inflammatory markers will be evaluated to investigate the potential anti-inflammatory effect of this treatment.
Exploratory Outcome -Interleukin-7 (IL-7) | Baseline to week 12 (+/- 7 days)
  Inflammatory markers will be evaluated to investigate the potential anti-inflammatory effect of this treatment.
Exploratory Outcome -Interleukin-8 (IL-8) | Baseline to week 12 (+/- 7 days)
  Inflammatory markers will be evaluated to investigate the potential anti-inflammatory effect of this treatment.
Exploratory Outcome -Interleukin-10 (IL-10) | Baseline to week 12 (+/- 7 days)
  Inflammatory markers will be evaluated to investigate the potential anti-inflammatory effect of this treatment.
Exploratory Outcome -Interleukin-10 receptor subunit alpha (IL-10RA) | Baseline to week 12 (+/- 7 days)
  Inflammatory markers will be evaluated to investigate the potential anti-inflammatory effect of this treatment.
Exploratory Outcome -Interleukin-10 receptor subunit beta (IL-10RB) | Baseline to week 12 (+/- 7 days)
  Inflammatory markers will be evaluated to investigate the potential anti-inflammatory effect of this treatment.
Exploratory Outcome -Interleukin-12 subunit beta (IL-12B) | Baseline to week 12 (+/- 7 days)
  Inflammatory markers will be evaluated to investigate the potential anti-inflammatory effect of this treatment.
Exploratory Outcome -Interleukin-13 (IL-13) | Baseline to week 12 (+/- 7 days)
  Inflammatory markers will be evaluated to investigate the potential anti-inflammatory effect of this treatment.
Exploratory Outcome -interleukin-15 receptor subunit alpha (IL-15RA) | Baseline to week 12 (+/- 7 days)
  Inflammatory markers will be evaluated to investigate the potential anti-inflammatory effect of this treatment.
Exploratory Outcome -Interleukin-17A (IL-17A) | Baseline to week 12 (+/- 7 days)
  Inflammatory markers will be evaluated to investigate the potential anti-inflammatory effect of this treatment.
Exploratory Outcome -Interleukin-17C (IL-17C) | Baseline to week 12 (+/- 7 days)
  Inflammatory markers will be evaluated to investigate the potential anti-inflammatory effect of this treatment.
Exploratory Outcome -Interleukin-20 (IL-20) | Baseline to week 12 (+/- 7 days)
  Inflammatory markers will be evaluated to investigate the potential anti-inflammatory effect of this treatment.
Exploratory Outcome -Interleukin-20 receptor subunit alpha (IL-20RA) | Baseline to week 12 (+/- 7 days)
  Inflammatory markers will be evaluated to investigate the potential anti-inflammatory effect of this treatment.
Exploratory Outcome -Interleukin-23 (IL-24) | Baseline to week 12 (+/- 7 days)
  Inflammatory markers will be evaluated to investigate the potential anti-inflammatory effect of this treatment.
Exploratory Outcome -Interleukin-22 receptor subunit alpha-1 (IL-22 RA1) | Baseline to week 12 (+/- 7 days)
  Inflammatory markers will be evaluated to investigate the potential anti-inflammatory effect of this treatment.
Exploratory Outcome -Interleukin-33 (IL-33) | Baseline to week 12 (+/- 7 days)
  Inflammatory markers will be evaluated to investigate the potential anti-inflammatory effect of this treatment.
Exploratory Outcome -Latency-associated peptide transforming growth factor beta 1 (LAP TGF-beta-1) | Baseline to week 12 (+/- 7 days)
  Inflammatory markers will be evaluated to investigate the potential anti-inflammatory effect of this treatment.
Exploratory Outcome -Leukemia inhibitory factor receptor (LIF-R) | Baseline to week 12 (+/- 7 days)
  Inflammatory markers will be evaluated to investigate the potential anti-inflammatory effect of this treatment.
Exploratory Outcome -Macrophage colony-stimulating factor 1 (CSF-1) | Baseline to week 12 (+/- 7 days)
  Inflammatory markers will be evaluated to investigate the potential anti-inflammatory effect of this treatment.
Exploratory Outcome -Macrophage inflammatory protein 1-alpha (MIP1 alpha) | Baseline to week 12 (+/- 7 days)
  Inflammatory markers will be evaluated to investigate the potential anti-inflammatory effect of this treatment.
Exploratory Outcome -Matrix metalloproteinase-1 (MMP-1) | Baseline to week 12 (+/- 7 days)
  Inflammatory markers will be evaluated to investigate the potential anti-inflammatory effect of this treatment.
Exploratory Outcome -Matrix metalloproteinase-10 (MMP-10) | Baseline to week 12 (+/- 7 days)
  Inflammatory markers will be evaluated to investigate the potential anti-inflammatory effect of this treatment.
Exploratory Outcome -Monocyte chemotactic protein 1 (MCP-1) | Baseline to week 12 (+/- 7 days)
  Inflammatory markers will be evaluated to investigate the potential anti-inflammatory effect of this treatment.
Exploratory Outcome -Monocyte chemotactic protein 2 (MCP-2) | Baseline to week 12 (+/- 7 days)
  Inflammatory markers will be evaluated to investigate the potential anti-inflammatory effect of this treatment.
Exploratory Outcome -Monocyte chemotactic protein 3 (MCP-3) | Baseline to week 12 (+/- 7 days)
  Inflammatory markers will be evaluated to investigate the potential anti-inflammatory effect of this treatment.
Exploratory Outcome -Monocyte chemotactic protein 4 (MCP-4) | Baseline to week 12 (+/- 7 days)
  Inflammatory markers will be evaluated to investigate the potential anti-inflammatory effect of this treatment.
Exploratory Outcome -Natural killer cell receptor 2B4 (CD244) | Baseline to week 12 (+/- 7 days)
  Inflammatory markers will be evaluated to investigate the potential anti-inflammatory effect of this treatment.
Exploratory Outcome -Neurotrophin-3 (NT-3) | Baseline to week 12 (+/- 7 days)
  Inflammatory markers will be evaluated to investigate the potential anti-inflammatory effect of this treatment.
Exploratory Outcome -Neurturin (NRTN) | Baseline to week 12 (+/- 7 days)
  Inflammatory markers will be evaluated to investigate the potential anti-inflammatory effect of this treatment.
Exploratory Outcome -Oncostatin-M (OSM) | Baseline to week 12 (+/- 7 days)
  Inflammatory markers will be evaluated to investigate the potential anti-inflammatory effect of this treatment.
Exploratory Outcome -Osteoprotegerin (OPG) | Baseline to week 12 (+/- 7 days)
  Inflammatory markers will be evaluated to investigate the potential anti-inflammatory effect of this treatment.
Exploratory Outcome -Programmed cell death 1 ligand 1 (PD-L1) | Baseline to week 12 (+/- 7 days)
  Inflammatory markers will be evaluated to investigate the potential anti-inflammatory effect of this treatment.
Exploratory Outcome -Protein S100-A12 (EN-RAGE) | Baseline to week 12 (+/- 7 days)
  Inflammatory markers will be evaluated to investigate the potential anti-inflammatory effect of this treatment.
Exploratory Outcome -Signaling lymphocytic activation molecule (SLAMF1) | Baseline to week 12 (+/- 7 days)
  Inflammatory markers will be evaluated to investigate the potential anti-inflammatory effect of this treatment.
Exploratory Outcome -SIR2-like protein 2 (SIRT2) | Baseline to week 12 (+/- 7 days)
  Inflammatory markers will be evaluated to investigate the potential anti-inflammatory effect of this treatment.
Exploratory Outcome -STAM-binding protein (STAMPB) | Baseline to week 12 (+/- 7 days)
  Inflammatory markers will be evaluated to investigate the potential anti-inflammatory effect of this treatment.
Exploratory Outcome -Stem cell factor (SCF) | Baseline to week 12 (+/- 7 days)
  Inflammatory markers will be evaluated to investigate the potential anti-inflammatory effect of this treatment.
Exploratory Outcome -Sulfotransferase 1A1 (ST1A1) | Baseline to week 12 (+/- 7 days)
  Inflammatory markers will be evaluated to investigate the potential anti-inflammatory effect of this treatment.
Exploratory Outcome -T-cell surface glycoprotein CD5 (CD5) | Baseline to week 12 (+/- 7 days)
  Inflammatory markers will be evaluated to investigate the potential anti-inflammatory effect of this treatment.
Exploratory Outcome -T cell surface glycoprotein CD6 isoform (CD6) | Baseline to week 12 (+/- 7 days)
  Inflammatory markers will be evaluated to investigate the potential anti-inflammatory effect of this treatment.
Exploratory Outcome -Thymic stromal lymphopoietin (TSLP) | Baseline to week 12 (+/- 7 days)
  Inflammatory markers will be evaluated to investigate the potential anti-inflammatory effect of this treatment.
Exploratory Outcome -TNF-beta (TNFB) | Baseline to week 12 (+/- 7 days)
  Inflammatory markers will be evaluated to investigate the potential anti-inflammatory effect of this treatment.
Exploratory Outcome -TNF-related activation-induced cytokine (TRANCE) | Baseline to week 12 (+/- 7 days)
  Inflammatory markers will be evaluated to investigate the potential anti-inflammatory effect of this treatment.
Exploratory Outcome -TNF-related apoptosis-inducing ligand (TRAIL) | Baseline to week 12 (+/- 7 days)
  Inflammatory markers will be evaluated to investigate the potential anti-inflammatory effect of this treatment.
Exploratory Outcome -Transforming growth factor alpha (TGF-alpha) | Baseline to week 12 (+/- 7 days)
  Inflammatory markers will be evaluated to investigate the potential anti-inflammatory effect of this treatment.
Exploratory Outcome -Tumor necrosis factor (ligand) superfamily, member 12 (TWEAK) | Baseline to week 12 (+/- 7 days)
  Inflammatory markers will be evaluated to investigate the potential anti-inflammatory effect of this treatment.
Exploratory Outcome -Tumor necrosis factor (TNF) | Baseline to week 12 (+/- 7 days)
  Inflammatory markers will be evaluated to investigate the potential anti-inflammatory effect of this treatment.
Exploratory Outcome -Tumor necrosis factor ligand superfamily member 14 (TNFSF14) | Baseline to week 12 (+/- 7 days)
  Inflammatory markers will be evaluated to investigate the potential anti-inflammatory effect of this treatment.
Exploratory Outcome -Tumor necrosis factor ligand superfamily member 9 (TNFSF9) | Baseline to week 12 (+/- 7 days)
  Inflammatory markers will be evaluated to investigate the potential anti-inflammatory effect of this treatment.
Exploratory Outcome -Urokinase-type plasminogen activator (uPA) | Baseline to week 12 (+/- 7 days)
  Inflammatory markers will be evaluated to investigate the potential anti-inflammatory effect of this treatment.
Exploratory Outcome -Vascular endothelial growth factor A (VEGF-A) | Baseline to week 12 (+/- 7 days)
  Inflammatory markers will be evaluated to investigate the potential anti-inflammatory effect of this treatment.
Exploratory Outcome - Carbamylated albumin | Baseline to week 12 (+/- 7 days)
  Carbamylated albumin will be obtained as an additional measure of renal function and metabolic status.
Exploratory Outcome - Glycosylatedalbumin | Baseline to week 12 (+/- 7 days)
  Glycosylated albumin will be obtained as a confirmatory marker of glucose control.

CONTACTS AND LOCATIONS:
Overall Officials: Noemi Lois, Study Chair — Belfast Health & Social Care Trust and Queen's University Belfast
Locations (1):
- Belfast Health & Social Care Trust, Belfast, Co Antrim, United Kingdom

IPD SHARING:
Plan to Share IPD: No